CLINICAL TRIAL: NCT01849042
Title: A Multicenter, Randomized, Open-label, Prospective Study to Estimate the add-on Effects of Memantine as Ebixa Oral Pump on Language in Moderate to Severe Alzheimer's Disease Patients Already Receiving Donepezil.
Brief Title: Effect of Memantine Oral Pump on Language in Patients With Probable Alzheimer's Disease
Acronym: ROMEO-AD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seol-Heui Han, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROMEO-AD 14394A
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Memantine; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- donepezil maintain group (Other): continue already taking same dose (5mg or 10mg per day) of donepezil who assigned donepezil group
  Interventions: Drug: donepezil
- add-on Ebixa oral pump group (Active Comparator): Ebixa dosage titration (5mg per day for 1week, then 10mg per day for 1week, then 15mg per day for 1week, then up to 20mg per day) add-on already taking donepezil (5mg or 10mg per day)
  Interventions: Drug: Ebixa; Drug: donepezil

INTERVENTIONS:
Drug: Ebixa — add-on of Ebixa oral pump already receiving donepezil with stable dosage
  Arms: add-on Ebixa oral pump group
Drug: donepezil

SUMMARY:
This study will evaluate the pharmacological efficacy on language capability and compliance with combination of new Ebixa oral pump and donepezil compared to donepezil only in patients with probable Alzheimer's disease. Primary objective is to evaluate the efficacy of memantine on language capability in moderate to severe Alzheimer's disease patients who are taking stable donepezil treatment.Secondary objectives are to evaluate the efficacy of maintain on cognitive function and disease progression with K-MMSE, NPI, ROSA, and SIB-short form in probable AD.

ELIGIBILITY:
Inclusion Criteria:

* probable Alzheimer's disease in accordance with NINCDS-ADRDA criteria
* MMSE score equal to or less than 20
* Brain CT or MRI scan performed within the past 12 months
* living or having regular visit at least three times a week from caregiver
* able to visit outpatient clinic and to perform cognitive function test
* already taking stable dose of donepezil for 3 months prior to screening
* subject and caregiver who signed informed consent

Exclusion Criteria:

* involved in another clinical trial within 4 weeks prior to screening
* severe or unstable disease: acute or severe asthma, unstable or severe cardiovascular disease, acute peptic ulcer,chronic renal failure
* bradycardia (pulse rate less than 50bpm), sick sinus syndrome
* any laboratory finding including cognitive impairments(vitamine B12 or folic acid, syphilis, thyroid disease)
* severe auditory or visual disturbance
* other degenerative disease or psychosis
* taken any drug used for the treatment of Alzheimer's disease or dementia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
AQ-WAB(Western aphasia battery) | Six months

SECONDARY OUTCOMES:
ROSA (Relevant Outcome Scale for Alzheimer's Disease) | six months

OTHER OUTCOMES:
SIB-short form | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk university medical center, Seoul, South Korea